CLINICAL TRIAL: NCT00568139
Title: Evaluierung Von Nebenwirkungen Einer Therapie Mit Mitotane Beim Nebennierenkarzinom- Evaluation of Side Effects of Mitotane in Adrenocortical Carcinoma
Brief Title: Evaluation of Side Effects of Mitotane
Status: Active, not recruiting | Type: Observational
Sponsor: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Martin Fassnacht, Head of Endocrinology, University of Wuerzburg
Other Study IDs: Wue-ACC-Mitotane
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2024-09

CONDITIONS: Adrenocortical Carcinoma
Keywords: adrenal cancer; mitotane (Lysodren); adverse events
MeSH Terms: conditions — Adrenocortical Carcinoma; Adrenal Gland Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum, plasma, and urine samples will be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mitotane: Patients with adrenocortical carcinoma treated with mitotane monotherapy

SUMMARY:
Mitotane is standard therapy in the treatment of adrenocortical carcinoma. However, many adverse effects are not well documented. Therefore, we are aiming at collecting data about adverse effects in patients treated with mitotane

ELIGIBILITY:
Inclusion Criteria:

* Adrenocortical carcinoma
* Treatment with mitotane monotherapy as first-line therapy (in adjuvant setting or advanced disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with adrenocortical carcinoma treated in our center or other ENSAT centers
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Documentation of adverse effects | from starting mitotane until discontinuation of mitotane (since this is very variable from patient to patient no specific number of days or weeks can be entered (standard therapy would be about 2 years) or start of additional other medical therapies
  Adverse effects will be documented using the NCI CTC AE v5.5

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fassnacht, MD, Principal Investigator — University of Wuerzburg
Locations (1):
- University Hospital, Würzburg, Germany